CLINICAL TRIAL: NCT04829994
Title: A Long Term Prospective Post Market Clinical Follow-up (PMCF) of the GYNECARE TVT EXACT® Continence System for the Treatment of Stress Urinary Incontinence
Brief Title: Post-Market Clinical Follow-Up onTVT EXACT® Continence System
Status: Active, not recruiting | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC_2020_05
Record Dates: First submitted 2021-03-17; First posted 2021-04-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stress Urinary Incontinence
Keywords: GYNECARE TVT EXACT® Continence System; SUI
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Intervention — There is no intervention, beyond necessary clinical care, in this study. The surgical procedures being performed within the study are identical to the surgical procedures subjects would receive as part of SOC.

SUMMARY:
The objective of this single arm, post market, clinical study is to evaluate the performance of Gynecare TVT EXACT® Continence System in women undergoing retropubic mid-urethral sling surgery for Stress Urinary Incontinence (SUI).

ELIGIBILITY:
Inclusion Criteria:

Subjects who satisfy all of the following criteria will be considered eligible for enrollment in this study:

1. Stress urinary incontinence symptoms
2. Stress urinary incontinence confirmed by diagnostic evaluation of a cough stress test
3. Female subjects ≥ 21 years of age requiring treatment of SUI
4. Desired surgical correction of stress urinary incontinence using a synthetic pubo-urethral vaginal sling
5. Planned surgery for primary stress incontinence without concomitant prolapse surgery
6. Patient able and willing to participate in follow-up
7. Subject or authorized representative has signed the approved informed consent

Exclusion Criteria:

Subjects meeting any of the following criteria will be considered not eligible for enrollment in this study:

1. Physical or psychological condition which would impair study participation or are unwilling or unable to participate in all required study visits and are unable to complete the questionnaires
2. Any pre-operative or intra-operative findings identified by the surgeon that may preclude the use of study product
3. History of previous synthetic, biologic or fascial pubo-urethral sling
4. Pregnancy or plans for future pregnancy
5. History of bleeding diathesis or current anti-coagulation therapy which cannot be suspended peri-operatively according to site's standard practice.
6. Current genitourinary fistula or urethral diverticulum
7. Reversible cause of incontinence (i.e. drug effect)
8. Contraindication to surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects ≥ 21 years of age
Study Population: Female subjects ≥ 21 years of age with a diagnosis of SUI, resulting from utrethral hypermobility and/or intrinsic sphincter deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2035-09-30 (Estimated); Study Completion 2036-02-28 (Estimated)

PRIMARY OUTCOMES:
Cough Stress Test (CST) Assessment Change | Post-surgery through study completion, approximately 5-10 yrs
  Objective cure of Stress Urinary Incontinence (SUI) (treatment success) sproximately 5-10 years after surgery, defined as a negative CST

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | Post-surgery through study completion, approximately 10 yrs
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline and post-surgery through study completion, approximately 10 yrs
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | Baseline and post-surgery through study, approximately 10 yrs completion
Wong-Baker FACES® Pain Rating Scale | Post-surgery through study completion, approximately 10 yrs
  To assess pain on a scale from 0 (no pain) to 10 (worst pain) related to study device or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.
Locations (8):
- United States (3):
  - Duke University, Durham, North Carolina
  - Institute for Female Pelvic Medicine, North Wales, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
- Ordensklinikum Linz, Linz, Austria
- Herlev Hospital, Hillerød, Denmark
- Hopital Jeanne de Flandres, Lille, France
- Universitatsklinikum Tubingen, Tübingen, Germany
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu